CLINICAL TRIAL: NCT03113487
Title: P53MVA and Pembrolizumab in Treating Patients With Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16448; NCI-2017-00555 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16448 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Platinum-Resistant Fallopian Tube Carcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma; Recurrent Platinum-Resistant Primary Peritoneal Carcinoma
MeSH Terms: interventions — MVAp53 vaccine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, p53MVA) (Experimental): Patients receive pembrolizumab IV over 30 minutes every 3 weeks and modified vaccinia virus ankara vaccine expressing p53 SC every 3 weeks for up to 3 vaccines. Cycles with pembrolizumab repeat every 3 weeks for up to 49 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Modified Vaccinia Virus Ankara Vaccine Expressing p53; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Modified Vaccinia Virus Ankara Vaccine Expressing p53 — Given SC
  Other Names: MVA-p53; MVA-p53 Vaccine; MVAp53 Vaccine; p53-MVA Vaccine; p53MVA
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well modified vaccinia virus ankara vaccine expressing p53 (p53MVA) and pembrolizumab work in treating patients with ovarian, primary peritoneal, or fallopian tube cancer that has come back (recurrent). Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving p53MVA and pembrolizumab together may work better in treating patients with ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess response rate (complete responses and partial responses) after treatment with p53MVA and pembrolizumab.

SECONDARY OBJECTIVE:

I. To assess median progression free survival (PFS), clinical benefit (complete response, partial response lasting > 6 months), overall survival (OS), safety and tolerability.

EXPLORATORY OBJECTIVE:

I. Evaluate if the CD8+ T cell signal exceeds that detected in the single agent p53MVA trial.

OUTLINE: This is a dose-escalation study of modified vaccinia virus ankara vaccine expressing p53.

Patients receive pembrolizumab intravenously (IV) over 30 minutes every 3 weeks and modified vaccinia virus ankara vaccine expressing p53 subcutaneously (SC) every 3 weeks for up to 3 vaccines. Cycles with pembrolizumab repeat every 3 weeks for up to 49 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1-3 weeks and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed diagnosis of epithelial ovarian, primary peritoneal or fallopian tube cancer will be enrolled in this study; patients must have experienced recurrence or progression within 6 months after completion of platinum based chemotherapy (by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria).
* A patient is eligible to participate if she is not pregnant, not breast-feeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) OR b.) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have measurable disease based on RECIST 1.1., or detectable disease; lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be greater than or equal to 10 mm when measured by computed tomography (CT), positron emission tomography (PET)/CT or magnetic resonance imaging (MRI); lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT, PET/CT, or MRI

  * Detectable disease in a patients is defined as one who does not have measurable disease, but has at least one of the following conditions:

    * Baseline values of CA-125 at least 2 x upper limit of normal (ULN)
    * Ascites and/ or pleural effusion attributed to tumor
    * Solid and/ or cystic abnormalities on radiographic imaging that do not meet modified RECIST criteria, immune-related response criteria (irRC) for target lesions
* Patients whose ovarian cancer recurs/progresses within 0-6 months following platinum-based chemotherapy have platinum resistant or refractory disease; these patients are not considered to benefit from additional platinum-based therapy and are treated with other sequential single agents; such patients are eligible for this trial
* Patients with documented disease recurrence/progression within 6-12 months of completing platinum-based therapy, are considered to have 'borderline' platinum sensitivity; these patients will not be eligible for this trial
* Patients who relapse more than 12 months after completion of platinum-based treatment are considered 'platinum sensitive' and will not be eligible for this trial, since they have a favorable (33-59%) chance of responding to further rounds of platinum based chemotherapy
* Patients with confirmed p53 mutation by molecular analysis and/or evidence of p53 overexpression by immunohistochemistry (>= 10% of cells within tumor staining positive) will be eligible; this will be assessed semi-quantitatively by a Clinical Laboratory Improvement Act (CLIA) approved pathology core pathologist, using CLIA approved mutational analysis or immuno-histochemistry techniques on formalin-fixed paraffin-embedded tissue; in the case of equivocal immunohistochemistry (IHC) results, p53 involvement may be confirmed by detection of p53 molecular analysis on tumor deoxyribonucleic acid (DNA); patients on whom molecular analysis of p53 mutations is already available, will not require IHC analysis; molecular analysis may be performed as an additional research procedure at the end of the study (distinct from eligibility determination) if the principal investigator (PI) deems it of scientific value and research funding is available to cover the cost; patients are not required to have PD-L1 positive ovarian tumors and PD-L1 testing is not mandatory on this study; however, we will collect the data on PD-L1 testing when available
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 (Karnofsky >= 60%) and a life expectancy of at least 3 months
* Up to 4 prior chemotherapy regimens for recurrent disease are allowed; adjuvant chemotherapy and maintenance Taxol after completion of six cycles of adjuvant carboplatin - Taxol will not be counted as a "prior chemotherapy regimen" for the purpose of this study; treatment with targeted agents or hormones would not be considered as a systemic chemotherapy regimen; eligible Patients are those with documented disease recurrence/progression within 0-6 months of completing platinum-based chemotherapy; patients should not have received any non-oncology, viral vaccines within 30 days prior to starting protocol treatment
* Absolute neutrophil count (ANC) >= 1500/uL (collected within 14 days prior to the start of study treatment)
* Platelets >= 100 000/uL (collected within 14 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (collected within 14 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 50 mL/min for participant with creatinine levels > 1.5 x institutional ULN (collected within 14 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (collected within 14 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (collected within 14 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (collected within 14 days prior to the start of study treatment)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (collected within 14 days prior to the start of study treatment)
* Left ventricle ejection fraction (LVEF) >= 55% (collected within 14 days prior to the start of study treatment)

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to study treatment start; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to treatment start

  * Note: participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline; participants with =< grade 2 neuropathy may be eligible
  * Note: if participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 3 weeks of start of study treatment; participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis; a 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment; Note: participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency (including organ grafts and human immunodeficiency virus [HIV]), or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug (exceptions: nasal corticosteroids, inhaled steroids, adrenal replacement steroids and steroid creams are allowed)
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years; Note: participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or any carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active CNS metastases and/or carcinomatous meningitis; participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV)
* Has active infection with hepatitis A (as determined by an acute hepatitis panel), a known history of hepatitis B (hepatitis B surface antigen [Ag] reactive), or active hepatitis C virus (qualitative hepatitis C virus [HCV] ribonucleic acid [RNA] detectable)
* Active TB (Bacillus tuberculosis) infection (as determined by Quantiferron Test)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Patients with a history of cardiac disease are excluded: myocardial infarction or arterial thromboembolic events within 6 months prior to baseline, severe or unstable angina, New York Heart Association Class III or IV disease, QTCB (corrected according to Bazett's formula) interval > 470 msec, serious uncontrolled hypertension (systolic > 150 and/or diastolic > 100 mm Hg); baseline electrocardiography, echocardiography and assessment of serum troponin (I) are included in the screening exams; subjects in whom these assays are abnormal (electrocardiogram [EKG] excluding 1st degree branch block, sinus brachycardia, sinus tachycardia or non-specific T wave changes, serum troponin >= grade 2) are ineligible
* Patients with a family history or Li-Fraumeni syndrome will not be eligible
* History of severe environmental allergies or allergy to egg proteins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2026-05-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Dellinger, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- p53MVA and Pembrolizumab: Patients received 5.6 × 10^8 pfu of p53MVA delivered as an intramuscular injection into the upper arm over the deltoid muscle followed by pembrolizumab 200 mg intravenously 30 minutes after vaccination. Both agents were given on day 1 of a 21-day cycle for three cycles, followed by single agent pembrolizumab 200 mg every 3 weeks up to 35 cycles (2 years total).
Period: Overall Study
Arm/Group | p53MVA and Pembrolizumab
Started | 29
Completed | 28
Not Completed | 1
Not completed — After cycle 1 sepsis was deemed present at baseline, so the patient was ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | p53MVA and Pembrolizumab
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: Years] | 64 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2
  Asian | 4
  Caucasian, Non-Hispanic | 15
  Hispanic | 7
Region of Enrollment [Number; unit: participants]
  United States | 28
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants]
  0: Fully active, with no performance restrictions | 13
  1: Restricted in strenuous activity, but fully ambulatory and able to carry out light work | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Complete or Partial Response
Description: Clinical response was assessed using the modified irRECIST criteria. Complete Response (CR) - Disappearance of all lesions, 2 consecutive observations, ≥ 4 wks apart; Partial Response (PR) - ≥50% decrease in tumor burden from baseline, 2 consecutive observations, ≥ 4 wks apart. Response = CR+PR.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | p53MVA and Pembrolizumab
Number analyzed (Participants) | 28
Participants | 3

2. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From initial treatment until progression or death. Progression is defined using Immune-related response criteria (irRECIST, irRC), as at least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 wks apart.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | p53MVA and Pembrolizumab
Number analyzed (Participants) | 28
Months | 1.8 [1.7 to 3.8]

3. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From the time of initial treatment until death from any cause.
Time Frame: From start of the treatment until death, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | p53MVA and Pembrolizumab
Number analyzed (Participants) | 28
Months | 15.1 [9.4 to 30.4]

4. Secondary Outcome: Clinical Benefit Rate
Description: Clinical response was assessed using the modified irRECIST criteria. Complete Response (CR) - Disappearance of all lesions, 2 consecutive observations, ≥ 4 wks apart; Partial Response (PR) - ≥50% decrease in tumor burden from baseline, 2 consecutive observations, ≥ 4 wks apart; Stable Disease (SD) - 50% decrease in tumor burden from baseline cannot be established, nor 25% increase compared with nadir. Clinical benefit = CR+PR+ stable disease [SD] > 6 months.
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | p53MVA and Pembrolizumab
Number analyzed (Participants) | 28
percentage of participants | 21.4

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment. Adverse events occurred over a period of 2 years and 4 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | p53MVA and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 17/28
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | p53MVA and Pembrolizumab (N=28)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | p53MVA and Pembrolizumab (N=28)
Anemia (Blood and lymphatic system disorders) | 10 (24)
Heart failure (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 5 (6)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 6 (21)
Hypothyroidism (Endocrine disorders) | 4 (10)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 10 (12)
Ascites (Gastrointestinal disorders) | 4 (4)
Bowel Urgency (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (20)
Diarrhea (Gastrointestinal disorders) | 8 (19)
Dry mouth (Gastrointestinal disorders) | 3 (29)
Dyspepsia (Gastrointestinal disorders) | 2 (5)
Dysphagia (Gastrointestinal disorders) | 1 (19)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (16)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (13)
gum tenderness (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 5 (7)
Edema limbs (General disorders) | 4 (9)
Fatigue (General disorders) | 15 (63)
Fever (General disorders) | 9 (17)
Flu like symptoms (General disorders) | 3 (3)
Injection site reaction (General disorders) | 27 (61)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (3)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4)
Wound infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time pr (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (11)
Alkaline phosphatase increased (Investigations) | 5 (10)
Aspartate aminotransferase increased (Investigations) | 4 (9)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 5 (6)
Lymphocyte count decreased (Investigations) | 3 (6)
Neutrophil count decreased (Investigations) | 2 (17)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (20)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (23)
Hyponatremia (Metabolism and nutrition disorders) | 9 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (38)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (39)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
hand cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Presyncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (5)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (18)
Insomnia (Psychiatric disorders) | 3 (5)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (12)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (7)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 7 (20)
Hypotension (Vascular disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03113487/Prot_SAP_000.pdf